CLINICAL TRIAL: NCT06175156
Title: The Application of Propofol and Remifentanil Mixed Solution for Controlled Sedation and Analgesia in Fiber Colonoscopy
Brief Title: Application of Propofol Mixed With Remifentanil in Fiber Colonoscopyand Analgesia in Fiber Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Handan First Hospital (Other)
Responsible Party: Principal Investigator, Yonghua Song, Director of Anesthesiology Department, Handan First Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-L-001
Record Dates: First submitted 2023-11-30; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Narcotism
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controlled analgesia/sedation (PCAS) group (Experimental): Each group of patients is required to open the right upper limb venous access as a routine, take the left side lying position, and continuously inhale oxygen with a mask at a flow rate of 8L/min, while connecting various monitoring devices. During the pre anesthesia assessment, explain in detail to the patient the usage of the self-control pump and confirm that each patient can master it. Firstly, connect the self-control analgesic pump with a loading dose of 3 ml. Then, continuously pump in a mixture of propofol and remifentanil at a speed of 0.1 ml/kg/h. After the loading dose is completed, the examination can begin. During the operation, press the self-control handle according to the patient's sensation. Each press can quickly push 1ml of the medication, with a locking time of 1 minute.
  Interventions: Procedure: Controlled analgesia/sedation
- Intravenous combined anesthesia group (Active Comparator): Each group of patients is required to open the right upper limb venous access as a routine, take the left side lying position, and continuously inhale oxygen with a mask at a flow rate of 8L/min, while connecting various monitoring devices. Intravenous slow infusion of fentanyl 1 μ G/kg, midazolam 0.02mg/kg, slowly administer propofol 0.8-1mg/kg after 2 minutes (time greater than 60 seconds), and start the examination when the patient's consciousness disappears and they do not respond. During the surgery, propofol is interrupted to maintain the auditory evoked potential index (AAI) between 30-40.
  Interventions: Procedure: Intravenous combined anesthesia

INTERVENTIONS:
Procedure: Controlled analgesia/sedation — During the pre anesthesia assessment, explain in detail to the patient the usage of the self-control pump and confirm that each patient can master it. Firstly, connect the self-control analgesic pump with a loading dose of 3 ml. Then, continuously pump in a mixture of propofol and remifentanil at a speed of 0.1 ml/kg/h. After the loading dose is completed, the examination can begin. During the operation, press the self-control handle according to the patient's sensation. Each press can quickly push 1ml of the medication, with a locking time of 1 minute
  Arms: Controlled analgesia/sedation (PCAS) group
Procedure: Intravenous combined anesthesia — Intravenous slow infusion of fentanyl 1 μ G/kg, midazolam 0.02mg/kg, slowly administer propofol 0.8-1mg/kg after 2 minutes (time greater than 60 seconds), and start the examination when the patient's consciousness disappears and they do not respond. During the surgery, propofol is interrupted to maintain the auditory evoked potential index (AAI) between 30-40.
  Arms: Intravenous combined anesthesia group

SUMMARY:
Fiber colonoscopy, as a terminal examination method for lower gastrointestinal diseases, often brings varying degrees of pain, discomfort, tension, and anxiety to patients. Therefore, currently in clinical practice, intravenous anesthesia is often chosen to reduce discomfort. At present, intravenous propofol and fentanyl are most widely used in clinical practice, but intravenous general anesthesia can lead to hemodynamic fluctuations and an increase in anesthesia related complications such as prolonged hospital stay after surgery. Propofol and remifentanil have the characteristics of fast onset, short duration of action, and rapid awakening. The purpose of this study is to observe the efficacy and adverse reactions of remifentanil combined with low-dose propofol in patient-controlled analgesia and sedation during colonoscopy, in order to explore the safety and effectiveness of this method.

DETAILED DESCRIPTION:
Fibercolonoscopy, as a terminal examination method for lower digestive tract diseases, often brings different degrees of pain and discomfort, tension and anxiety to patients. Therefore, at present, intravenous anesthesia is often used in clinical practice to reduce discomfort, and intravenous propofol combined with fentanyl is the most widely used in clinical practice. But intravenous general anesthesia can lead to hemodynamic fluctuations and an increase in anesthesiation-related complications such as longer stays in the hospital after surgery. Complications related to sedation and analgesia have attracted increasing attention in recent years. Studies have shown that most of the adverse events in endoscopy are related to the sedation and analgesia drugs used. With the successful application of patient-controlled analgesia (PCA) in the field of postoperative analgesia, this technique has also been used in the sedation and analgesia of gastroenteroscopy in recent years. Propofol has the characteristics of quick action, short time of action and rapid recovery, so it is very suitable for the anesthesia and sedation of painless abortion and painless gastroenteroscopy. Remifentanil, as an opioid μ receptor agonist, is easily hydrolyzed rapidly by non-specific esterases in plasma and tissues due to the ester bond contained in its chemical structure. Therefore, it has unique pharmacokinetic characteristics such as rapid intravenous injection, small volume of distribution, rapid clearance after drug withdrawal, no accumulation, metabolism is not affected by liver and kidney function, and has been widely used in various surgeries in recent years, especially in the anesthesia of short surgeries.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) Grade I - II;
2. Age 18-75 years old;
3. Body mass index (BMI) <25㎏/㎡;
4. no mental and nervous system diseases;

Exclusion Criteria:

1. Refusal to cooperate or difficulty communicating;
2. History of drug allergy;
3. Long-term alcoholism and dependence on stabilizing and opioid drugs;
4. Patients with past history of intestinal surgery or past difficulty in endoscopic surgery;
5. People with hearing impairment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Auditory evoked potential | through study completion，an average of 2 hours
  The auditory evoked potential (AEPI) is a reactive electrical activity of the brain generated by auditory stimuli, reflecting the entire electrical activity from the cochlea to the cerebral cortex.Before taking anesthesia, check Record the AEPI values at 5 time points before anesthesia, at the beginning of the examination, during endoscopy to the splenic curvature, ileocecal region, and at the end of the examination.

SECONDARY OUTCOMES:
The time from after surgery to OAA/S score reached 5 and Aldrete score reached 9 | through study completion，an average of 2 hours
  Evaluation and score were performed every minute after operation The time from surgery to OAA/S score of 5 and Aldrete score of 9 were recorded

OTHER OUTCOMES:
Intraoperative noninvasive blood pressure (MAP) | through study completion，an average of 2 hours
  Intraoperative noninvasive blood pressure (MAP) were monitored by nasal catheterization (ETCO2)
Pulse oximetry were monitored continuously Saturation (SPO2) | through study completion，an average of 2 hours
  pulse oximetry were monitored continuously Saturation (SPO2)were monitored by nasal catheterization (ETCO2)

CONTACTS AND LOCATIONS:
Locations (1):
- Handan First Hospital, Handan, Hebei, China

IPD SHARING:
Plan to Share IPD: No